CLINICAL TRIAL: NCT02678754
Title: A Registry of Caris Life Sciences® Molecular Intelligence™ Service (Biomarker Assessment Results) Intended for Correlation With Cancer Clinical Outcomes
Brief Title: Caris Molecular Intelligence Registry
Acronym: CMIR
Status: Terminated | Type: Observational
Why Stopped: Business decision to move away from this study
Sponsor: Caris Science, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TCREG-001-00-V2-1209
Record Dates: First submitted 2016-01-13; First posted 2016-02-10 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Solid Tumors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No intervention required, purely observational

SUMMARY:
This data collection Registry is a multi-center, observational outcomes Database designed to collect data on the demographics, presentation, diagnosis, treatment, resource use, quality of life and outcomes of subjects utilizing Caris Molecular Intelligence™ Services for treatment of solid tumor cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years, and
* Solid Tumor analyzed by Caris Molecular Intelligence™ Service Profile(s) and/or Caris Next-Generation Sequencing

Exclusion Criteria:

* Individual test orders; defined as single biomarker assessment
* Due to the complexity of state and federal requirements governing the participation of prisoners in research, prisoner-patients shall not be approached for participation in the Registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients seen within a physician practice participating in the Registry are potential candidates if they meet the eligibility criteria requirements
Sampling Method: Probability Sample
Enrollment: 4981 (Actual)
Dates: Start 2010-02; Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Documentation of the frequency of specific clinical events in relation to risk factors, diagnosis and treatments provided. | 5 years per patient